CLINICAL TRIAL: NCT03414866
Title: Thoraflex Hybrid Post-Market Study
Acronym: THOR
Status: Active, not recruiting | Type: Observational
Sponsor: Vascutek Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: THOR-001
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Acute Aortic Dissection; Aortic Rupture; Penetrating Aortic Ulcer; Aortic Dissection; Aortic Aneurysm, Thoracic
Keywords: Thoracic Aorta; Dissection; Aneurysm; Frozen Elephant Trunk
MeSH Terms: conditions — Aortic Rupture; Penetrating Atherosclerotic Ulcer; Aortic Dissection; Aortic Aneurysm, Thoracic; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Acute thoracic aortic syndrome: 60 patients, standard of care (non-interventional) EQ-5D-5L QOL Questionnaire
  Interventions: Behavioral: EQ-5D-5L QOL questionnaire
- Subacute/chronic dissection of the aorta: 60 patients, standard of care (non-interventional) EQ-5D-5L QOL Questionnaire
  Interventions: Behavioral: EQ-5D-5L QOL questionnaire
- Aortic aneurysm: 60 patients, standard of care (non-interventional) EQ-5D-5L QOL Questionnaire
  Interventions: Behavioral: EQ-5D-5L QOL questionnaire

INTERVENTIONS:
Behavioral: EQ-5D-5L QOL questionnaire — Written questionnaire

SUMMARY:
This is a global, prospective non-interventional, multi-centre, post-market study of the Vascutek Thoraflex™ Hybrid system in patients with acute thoracic aortic syndrome, subacute/chronic dissection of the aorta and aortic aneurysm.

DETAILED DESCRIPTION:
Aortic arch pathologies are rare, but pose significant challenges for treatment involving open surgical or endovascular repair.

In 1983 the Elephant Trunk technique was introduced and has greatly facilitated the management of patients with extensive thoracic aortic disease.

In recent years, this traditional open surgery has been combined with thoracic endovascular repair (TEVAR) and this is known as the 'hybrid' approach. Hybrid repairs, consisting of an open surgical repair combined with endovascular techniques.

Further advancement in the types of prosthesis available has resulted in the evolution of the conventional ET technique into the frozen elephant trunk (FET) technique. This utilises devices that incorporate both a traditional dacron graft (for open surgical treatment of the aortic arch) and a stented graft portion (for treatment of the descending thoracic aorta). The stented portion of the graft is introduced via an antegrade approach through the transected arch. The FET technique is now commonly used to treat patients with extensive thoracic or thoraco-abdominal aortic disease.

Vascutek Ltd has developed the Thoraflex™ Hybrid Device (Plexus™ 4 and Ante-Flo™) for the repair or replacement of damaged or diseased vessels of the ascending aorta, aortic arch and descending thoracic aorta in cases of aneurysm and/or dissection. The Thoraflex™ Hybrid Device is one of the commercially available frozen elephant trunk prosthesis.

Over 3000 Thoraflex™ Hybrid Devices have been sold and the current study seeks to provide further evidence of the continuing safety and effectiveness of the device.

ELIGIBILITY:
Inclusion Criteria:

* Patient is aged 18 years or over on date of consent
* Patient is willing and able to comply with all study procedures and study visits
* Patient or their legally authorised representative (LAR) has given written informed consent to participate in study. For emergency patients only, retrospective consent is permissible
* Patient satisfies the inclusion criteria for one of the following categories:

A - Patient has acute thoracic aortic syndrome or B - Patient has subacute/ chronic dissection of the aorta or C - Patient has an aortic aneurysm (including connective tissue disorders)

A. Patients with acute thoracic aortic syndrome:

Patient has acute thoracic aortic syndrome and requires repair or replacement of damaged or diseased vessels of the aortic arch (with or without involvement of the ascending aorta), and the descending aorta requires replacement, or, in the opinion of the investigator, the patient would derive clinical benefit from prophylactic treatment of the descending aorta. This includes patients with acute dissections, rupture of the aorta or PAU.

B. Patients with subacute/chronic dissection of the aorta:

* Patient requires repair or replacement of damaged or diseased vessels of the aortic arch and descending aorta with or without involvement of the ascending aorta due to subacute/chronic dissection.

And patient satisfies one or more of the following criteria:

* Patient has aortic sinus, or ascending aorta, or aortic arch, or descending aorta diameter ≥5.5cm (including if asymptomatic) or
* Patient has aorta diameter <5.5cm and growth rate ≥0.5cm/year (including if asymptomatic) or
* Patient has ascending aorta diameter ≥4.5cm and requires valve repair or replacement

C. Patients with an aortic aneurysm (including connective tissue disorders):

* Patient requires repair or replacement of damaged or diseased vessels of the aortic arch and descending aorta with or without involvement of the ascending aorta

And patient satisfies one or more of the following criteria:

* Patient has aortic sinus, or ascending aorta, or aortic arch, or descending aorta diameter ≥5.5cm (including if asymptomatic) or
* Patient has aorta diameter <5.5cm and growth rate ≥0.5cm/year (including if asymptomatic) or
* Patient has ascending aorta diameter ≥4.5cm and requires valve repair or replacement.

or

* Patient has Marfan syndrome or other genetically mediated disorders with aortic sinus, or ascending aorta, or arch diameter ≥4.5cm, or, the ratio of the maximal ascending or aortic root area (Π r2) in cm2 divided by the patient's height in meters exceeds 10

Exclusion Criteria:

* Patient is unfit for open surgical repair involving circulatory arrest
* Patient has known sensitivity to polyester, nitinol or materials of bovine origin
* Patient has active endocarditis or an active infective disorder of the aorta
* Patient has an active systemic infection that, in the opinion of the investigator, would compromise the outcome of the surgical procedure
* Patient is enrolled in another active study and has received an investigational product (device, pharmaceutical or biologic) within 6 months prior to the date of the implant or has not reached the primary endpoint of the study, which in the opinion of the Investigator will impact on this study
* Patient has an uncorrectable bleeding anomaly
* Patient has renal failure (defined as dialysis dependent)
* Patient has known sensitivity to radiopaque contrast agents that cannot be adequately pre-treated
* Patient has a co-morbidity causing expected survival to be less than 1 year
* Patient has any other medical, social or psychological problems that in the opinion of the investigator preclude them from receiving this treatment and the procedures and evaluations pre and post procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients with acute thoracic aortic syndrome, including: acute dissection, aortic rupture and penetrating aortic ulcer (PAU)
  60 patients with a subacute/chronic dissection of the aorta
  60 patients with an aortic aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Freedom from Major Adverse Event | 1 year post-procedure
  The primary endpoint will be freedom from the following composite Major Adverse Event (MAE): permanent stroke , permanent paraplegia/paraparesis, unanticipated aortic related re-operation (excluding re-operation for bleeding) and aortic related mortality

CONTACTS AND LOCATIONS:
Overall Officials: Malakh Shrestha, Prof. Dr., Principal Investigator — Hannover Medical School
Locations (7):
- Canada (3):
  - London Health Sciences Centre, University Hospital, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
- Germany (2):
  - University of Freiburg, Freiburg im Breisgau
  - Hannover Medical School, Hanover
- Policlinico S.Orsola-Malpighi, Bologna, Italy
- St Antonious Hospital, Nieuwegein, Netherlands